CLINICAL TRIAL: NCT03954327
Title: Randomized Controlled Trail (RCT) of Emtricitabine, Tenofovir Disoproxil and Raltegravir for Patients With Primary Biliary Cholangitis Unresponsive to Ursodeoxycholic Acid (UDCA)
Brief Title: Combination Antiretroviral Therapy (cART) for PBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00082571
Record Dates: First submitted 2019-05-07; First posted 2019-05-17 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emtricitabine (FTC)/Tenofovir Disoproxil (TDF) & Raltegravir (Experimental): one Emtricitabine 200mg and Tenofovir Disoproxil 300mg tablet two Raltegravir 600mg tablets
  Interventions: Drug: Emtricitabine (FTC)/Tenofovir Disoproxil (TDF); Drug: Raltegravir
- Placebo (Placebo Comparator): Identical tablets resembling one Emtricitabine 200mg and Tenofovir Disoproxil 300mg tablet two Raltegravir 600mg tablets
  Interventions: Drug: Placebo Oral Capsule [CEBOCAP]

INTERVENTIONS:
Drug: Emtricitabine (FTC)/Tenofovir Disoproxil (TDF) — Emtricitabine (FTC) 200 mg/Tenofovir Disoproxil (TDF) 300 mg by mouth once per day
  Other Names: Truvada
  Arms: Emtricitabine (FTC)/Tenofovir Disoproxil (TDF) & Raltegravir
Drug: Raltegravir — Raltegravir (RTF) 600 mg two tablets by mouth once per day
  Other Names: Isentress
  Arms: Emtricitabine (FTC)/Tenofovir Disoproxil (TDF) & Raltegravir
Drug: Placebo Oral Capsule [CEBOCAP] — Two capsules identical to Raltegravir and one capsule identical to Truvada with no active ingredients by mouth once per day
  Other Names: placebo
  Arms: Placebo

SUMMARY:
Placebo Controlled, double-blind randomized controlled trial (RCT) with 12 months Tenofovir Disoproxil and Raltegravir for primary biliary cholangitis (PBC) patients unresponsive to Ursodeoxycholic Acid (UDCA). Placebo patients will be offered 12 months open label therapy at unblinding. All patients will be offered an additional 12 months open label therapy. Observational, open label study will be performed in parallel using Emtricitabine (FTC)/Tenofovir Disoproxil (TDF) & Raltegravir in liver transplant recipients meeting all entry criteria except for use of immunosuppression.

DETAILED DESCRIPTION:
Primary endpoint:

Change in mean percentage of alkaline phosphatase (ALP) reduction in cART vs. placebo at 6 and 12 months.

Secondary endpoints:

1. Serum biochemistries bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and gamma-glutamyltransferase (GGT) will be studied as continuous variables.
2. Composite endpoint used for the POISE study [A Placebo-Controlled Trial of Obeticholic Acid in Primary Biliary Cholangitis]: (i) reduction of ALP to < 1.67 upper limit of normal, (ii) normalization of bilirubin within upper limit of normal (ULN) and (iii) reduction of ALP by > 15% at 6 and 12 months.
3. Symptomatic evaluation performed using the PBC-40 to assess five symptom domains relating to fatigue, itch, cognitive symptoms, social and emotional symptoms, and other symptoms.
4. Histological change in grade and stage of PBC using the Nakanuma scoring system for a subgroup of patients undergoing liver biopsy [liver biopsy not compulsory for study].
5. Serial human betaretrovirus measurement in peripheral blood and cellular immune response to viral peptides.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old of either sex,
* Anti-mitochondrial antibody +ve or liver histology compatible with PBC,
* stable UDCA dose of 13-15 mg/kg for > 12 months or intolerant to UDCA,
* ALP at least 1.67 x ULN or abnormal bilirubin less than 2x ULN
* able to read and sign informed consent form.

Exclusion Criteria:

* subjects with baseline total bilirubin > 2 x ULN,(patients meeting inclusion criteria stabilized on second line therapies including obeticholic acid or bezafibrate over 12 months or more may be enrolled).
* use of non-standard or experimental therapy within the last 6 months,
* advanced liver disease: INR > 1.2 ULN, Albumin < 35 g/L lower limit of normal, platelets < 120,000/microL unless varices with risk of bleeding excluded by endoscopy within the last 6 months, Childs Pugh class B or C cirrhosis, presence of grade 2 varices or previous variceal hemorrhage, encephalopathy, ascites or need for liver transplantation within the next two years;
* secondary diagnosis such as HIV, viral hepatitis, drug induced liver injury, extrahepatic biliary obstruction, primary sclerosing cholangitis, metabolic liver - regular use of > 30g alcohol/day in the last year;
* a predicted survival of less than 3 years from malignant or other life threatening disease;
* hepatic mass consistent with hepatocellular carcinoma ;
* previous allergic reaction to study medications;
* Glomerular Filtration Rate less than < 30 mL/min as measured Cockcroft-Gault formula;
* pregnancy, breast-feeding or pre-menopausal patients not using contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Change in alkaline phosphatase levels | 12 months
  Mean changes in alkaline phosphatase levels after 12 months treatment with combination antiretroviral therapy or placebo.

SECONDARY OUTCOMES:
Serial changes in alkaline phosphatase | Evaluation baseline, 3 months, 6 months and end of RCT; then 3 months, 6 monthly to end of open label therapy]
  Serial changes in alkaline phosphatase levels with combination antiretroviral therapy or placebo.
Serial changes in ALT | Evaluation baseline, 3 months, 6 months and end of RCT; then 3 months, 6 monthly to end of open label therapy]
  Serial changes in ALT levels with combination antiretroviral therapy or placebo.
Serial changes in bilirubin | Evaluation baseline, 3 months, 6 months and end of RCT; then 3 months, 6 monthly to end of open label therapy]
  Serial changes in bilirubin levels with combination antiretroviral therapy or placebo.
Achievement of the composite biochemistry endpoint | 6 and 12 months
  (i) reduction of ALP to < 1.67 upper limit of normal, (ii) normalization of bilirubin within ULN and (iii) reduction of ALP by > 15%
Human Betaretrovirus load in peripheral blood | Evaluation baseline, 3 months, 6 months and end of RCT; then 3 months, 6 monthly to end of open label therapy
  Quantification of Human Betaretrovirus DNA or RNA levels in peripheral blood measured by Quantigene or polymerase chain reaction with therapy or placebo.
Interferon gamma release to Human Betaretrovirus peptide stimulation | Evaluation at baseline, 6 months and end of RCT; then 6 monthly to end of open label therapy
  Concentration of interferon gamma released from peripheral blood mononuclear cells stimulated by Human Betaretrovirus peptides in vitro in response to treatment or placebo.
Liver histology | Pretreatment biopsy and 24 month biopsy after initiation of study therapy
  Liver histology will be measured in a scale for staging and grading disease using the Nakanuma scoring system. Scores for fibrosis, bile duct loss, and chronic cholestasis will be combined for staging: stage 1, total score of 0; stage 2, score 1-3; stage 3, score 4-6; and stage 4, score 7-9. Cholangitis activity and hepatitis activity will be graded as 0-3, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Mason, MD, Principal Investigator — University of Alberta
Locations (6):
- Canada (6):
  - University of Alberta, Edmonton, Alberta
  - St Paul's Hospital, University of British Columbia, Vancouver, British Columbia
  - Vancouver General Hospital, University of Brittish Columbia, Vancouver, British Columbia
  - University of Toronto, Toronto, Ontario
  - University of Montreal, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No